CLINICAL TRIAL: NCT00633555
Title: A Randomized Controlled Trial of Microdose Leuprolide Protocol vs. Luteal Phase Ganirelix Protocol in Predicted Low Responders
Brief Title: A Comparison of the Microdose Leuprolide Protocol vs. Luteal Phase Ganirelix Protocol in Women Who Are or Who Are Predicted to be Low Responders
Acronym: LR
Status: Completed | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Other Study IDs: 06-198-2; CARS-06-198
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who have undergone in vitro fertilization (IVF) and produced four or less follicles or had four or less oocytes (eggs) retrieved are often referred to as poor responders. We will refer to these patients from this point forward as "low responders" to avoid using a potentially offensive label. We are currently using 2 different IVF medication protocols in our practice to treat low responder patients with infertility: the "Microdose Leuprolide" protocol and the "Luteal Phase Ganirelix" protocol. We would like to conduct a randomized-controlled trial and randomize patients to one treatment group or the other to determine which medication protocol is more effective in treating infertility in this group of patients.

DETAILED DESCRIPTION:
Women who demonstrate a suboptimal response to controlled ovarian hyperstimulation (COH) are a challenge to treat with assisted reproductive technologies such as in vitro fertilization (IVF). Such patients are often referred to clinically and in the medical literature as poor responders. A variety of different protocols have been studied and used to treat these patients. One protocol used to treat poor responders is the microdose leuprolide flare protocol 1,2. This widely-used protocol was first described in 1997 by Schoolcraft et al. 1 The microdose leuprolide flare protocol is so named because the administration of a gonadotropin-releasing hormone agonist (GnRH-a) in the early follicular phase causes an initial rise in endogenous gonadotropins called a "flare" before it causes downregulation and suppression of gonadotropins. Use of oral contraceptive pills (OCPs) in the preceding cycle prevents corpus luteum formation which could be supported by exogenous GnRH-a in the subsequent cycle. The microdose leuprolide flare protocol has been shown to be a safe and effective protocol which may lead to decreased cycle cancellation rates and increased clinical and ongoing pregnancy rates in poor responders 2,3.

The development of GnRH antagonists led to additional treatment options for poor responders 4. With GnRH antagonist use, suppression in the early follicular phase may be avoided. The GnRH antagonist is then added in the late follicular phase to prevent an LH surge. This protocol may enable a poor responder to recruit more follicles in the early follicular phase and thus have a more optimal response to stimulation. A randomized-controlled multicenter trial comparing the GnRH antagonist ganirelix to a GnRH agonist (Buserelin, intranasal preparation) in patients using recombinant FSH (rFSH) showed that ganirelix was safe and well-tolerated 5. They found that the mean duration of stimulation was 1 day shorter in the ganirelix group and that this group used significantly less rFSH. A randomized-controlled clinical trial of poor responders comparing the use of ganirelix to microdose leuprolide acetate (GnRH-a) in patients undergoing COH for IVF found that the outcomes were similar in both groups 6. There were no differences in total number of days of stimulation, amount of rFSH used, peak estradiol levels, number of oocytes retrieved, fertilization rate, implantation rate, or pregnancy rate. However, this study was limited by a small sample size. Another randomized-controlled trial by Akman et al. 7 compared the use of microdose leuprolide to GnRH antagonist (Cetrotide) in poor responders undergoing IVF. They found no difference in implantation rates and clinical pregnancy rates but were also limited by a small sample size.

In IVF cycles, poor responders often develop a dominant follicle and multiple small follicles rather than multiple large follicles which is the goal of such treatment. In such cases, the IVF cycle is often cancelled. The physiology behind such asynchronous follicular growth during COH is poorly understood. Such discrepant growth may be the result of size differences in early antral follicles 8. It is also possible that the premature FSH elevation that occurs in the late luteal phase of the menstrual cycle plays a role in this process 9. FSH prevents follicular atresia at the end of the luteal phase10. Some follicles are intrinsically more sensitive to FSH and able to respond to low levels of this hormone than others. Given the fact that larger follicles are often more FSH-responsive than small follicles, it makes sense that exogenous gonadotropins may lead to worsening follicular asynchrony during COH 11.

It has recently been shown that the use of estradiol in the luteal phase of the preceding menstrual cycle may facilitate growth of follicles in a coordinated fashion 8, 11. Fanchin et al.11 prospectively studied 90 women who were undergoing IVF cycles using GnRH antagonists and randomly assigned them to receive either 4 mg of oral micronized estradiol from cycle day 20 until day 2 of the next cycle or to serve as controls and receive no estradiol treatment. They found that the group that received estradiol had significantly smaller follicles on day 8 of their cycle and had less of a discrepancy in follicle size.. The group that received estradiol also had more follicles that were 16 mm or greater, more mature oocytes, and more embryos than the control group. The clinical pregnancy rate was greater in the estradiol group although this finding was not statistically significant (34 vs. 25%).

Recently, GnRH antagonists have also been shown to coordinate follicular size and subsequent growth when used in the luteal phase of the preceding menstrual cycle 12,13. Dragesic et al. 13 developed a novel protocol for poor responders which incorporated both transdermal estradiol (E2)and GnRH antagonist use in the luteal phase, followed by gonadotropin stimulation in the follicular phase and the addition of a GnRH antagonist in the late follicular phase. From this point on, this protocol will be referred to as the Luteal Phase Ganirelix (LPG) Protocol. During the LPG protocol, subjects applied a 0.1 mg transdermal estradiol patch on the 10th day after the LH surge and replaced this patch with a fresh 0.1 mg patch every other day. On the second day of patch use, subjects began taking daily ganirelix acetate 0.25 mg subcutaneously for 3 days. Subjects presented for ultrasound on day 2 of menses for FSH, LH, E2 and an ultrasound and stimulation was started per protocol with gonadotropins (rFSH and human menopausal gonadotropin (HMG)). Ganirelix was started when a 13mm follicle was measured on ultrasound, E2 exceeded 300 pg/mL, or on cycle day 7. Human chorionic gonadotropin (hCG) was given for final oocyte maturation and oocyte retrieval was performed 35-36 hours later. All embryo transfers were performed 72 hours after oocyte retrieval. This retrospective study of 68 subjects compared their responses to the LPG protocol with their responses to a prior IVF cycle protocol, which included microdose leuprolide, low-dose leuprolide, and coflare protocols. They found that when patients used the LPG Protocol they had significantly lower cycle cancellation rates, more oocytes retrieved, more mature oocytes, more normally fertilized oocytes, and more embryos available for transfer compared to their prior cycles. Patients did use more gonadotropins during the LPG protocol and had more days of stimulation, although the latter was not statistically significant.

Our goal in our proposed study is to determine whether the Microdose Leuprolide and LPG Protocols are equally efficacious in treating poor responders.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 21-44 undergoing IVF for infertility
* Prior IVF cycle with poor response (≤4 follicles on ultrasound,≤ 4 oocytes retrieved, peak estradiol <1000 pg/mL, prior IVF cycle cancelled for poor response)

OR

* Predicted poor response (age >40, basal FSH ≥10 mIU/mL, prior poor response to gonadotropin (peak estradiol <500 pg/mL))

Exclusion Criteria:

* Medical contraindications for oral contraceptive pills, injectable gonadotropin medications, estradiol, or progesterone in oil use.
* Medical contraindications to pregnancy
* Prior IVF cycle with Microdose Protocol or Luteal Phase Ganirelix Protocol

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women ages 21-44 who are currently undergoing In Vitro Fertilization treatment at our center.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 4-6 weeks

SECONDARY OUTCOMES:
Number of oocytes retrieved | 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Nulsen, MD, Principal Investigator — The Center for Advanced Reproductive Services, P.C.